CLINICAL TRIAL: NCT00293410
Title: Phase I Dose-Escalation Trial of Clofarabine Followed by Escalating Doses of Fractionated Cyclophosphamide in Adults and Children With Relapsed or Refractory Acute Leukemias
Brief Title: Clofarabine and Cyclophosphamide in Treating Patients With Relapsed or Refractory Acute Leukemia, Chronic Myelogenous Leukemia, or Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: J0561 CDR0000456431; P30CA006973 (NIH); JHOC-J0561; JHOC-00000845
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic/Myeloproliferative Diseases
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; accelerated phase chronic myelogenous leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; acute undifferentiated leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute promyelocytic leukemia (M3); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute basophilic leukemia; childhood acute monocytic leukemia (M5b); childhood acute eosinophilic leukemia; childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute minimally differentiated myeloid leukemia (M0); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Blast Crisis; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Clofarabine; Cyclophosphamide

INTERVENTIONS:
Drug: clofarabine
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine and cyclophosphamide in treating patients with relapsed or refractory acute leukemia, chronic myelogenous leukemia, or myeloproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and tolerability of administering clofarabine and fractionated cyclophosphamide in patients with relapsed or refractory acute leukemia, chronic myelogenous leukemia, or high-risk myeloproliferative disorders
* Determine the maximum tolerated dose of clofarabine and fractionated cyclophosphamide in these patients.
* Determine the toxic effects of these drugs in these patients.

Secondary

* Obtain preliminary data of biologic and pharmacodynamic effects of this regimen on marrow and circulating leukemic blasts in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to age (adult vs child).

Patients receive cyclophosphamide IV over 2 hours on day 0. Patients then receive clofarabine IV over 2 hours and cyclophosphamide IV over 2 hours on days 1-3 and 8-10. Treatment with clofarabine and cyclophosphamide repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of clofarabine and cyclophosphamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 10 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leukemia or myeloproliferative disorders, including 1 of the following:

  * Acute myeloid leukemia (AML) of any subtype

    * Treatment-related AML OR AML evolving from myeloproliferative disorders (MPD) or transformed from myelodysplastic syndrome
  * Acute lymphocytic leukemia
  * Acute progranulocytic leukemia

    * Must not be eligible for arsenic or retinoic acid therapy
  * Chronic myelogenous leukemia in accelerated phase or blast crisis
  * High-risk MPD, including any of the following:

    * Myelofibrosis
    * Chronic myelomonocytic leukemia with 5%-19% blasts
    * Relapsed or refractory juvenile myelomonocytic leukemia
* Relapsed and/or refractory disease with progressive disease since last therapy

  * No more than 3 prior induction regimens with cytotoxic agents for adults
  * Must be in second relapse for patients < 21 years of age

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2 (for adults) OR Lansky 50-100% (for pediatric patients)
* Bilirubin ≤ 1.5 mg/dL (may be elevated due to hemolysis in adult patients)
* AST and ALT ≤ 5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL (for adults)
* Normal renal function (for pediatric patients)
* Cardiac function normal as measured by MUGA scan or echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 6 months after completion of study treatment
* HIV negative
* No active graft-versus-host disease ≥ grade 2
* No active, uncontrolled infection
* No fever
* No unstable CT scans of the lungs, sinuses, or abdomen within the past 4 weeks
* No arrhythmias (other than atrial flutter or fibrillation) requiring medication
* No dyspnea at rest or with minimal exertion
* No uncontrolled congestive heart failure
* No myocardial infarction within the past 3 months
* No history of severe coronary artery disease
* No other significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance or interfere with consent, study participation, follow up, or interpretation of study results

PRIOR CONCURRENT THERAPY:

* Must have recovered from all acute toxic effects from prior treatment
* More than 30 days since prior investigational cytotoxic agents
* At least 3 days since prior azacitidine, thalidomide, hydroxyurea, imatinib mesylate, or interferon
* At least 1 week since prior growth factors except epoetin alfa
* More than 3 weeks since any other prior anticancer therapy
* No concurrent chemotherapy, radiotherapy, or immunotherapy
* No other concurrent anticancer investigational or commercial agents
* No routine prophylactic use of a colony-stimulating factor (filgrastim [G-CSF] or sargramostim [GM-CSF])

  * Therapeutic use of colony-stimulating factors may be considered at the discretion of the investigator
* No prolonged use of corticosteroids to prevent or treat emesis or as a chemotherapeutic agent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Karp JE, Ricklis RM, Balakrishnan K, Briel J, Greer J, Gore SD, Smith BD, McDevitt MA, Carraway H, Levis MJ, Gandhi V. A phase 1 clinical-laboratory study of clofarabine followed by cyclophosphamide for adults with refractory acute leukemias. Blood. 2007 Sep 15;110(6):1762-9. doi: 10.1182/blood-2007-03-081364. Epub 2007 Jun 11. PMID 17562873